CLINICAL TRIAL: NCT01274832
Title: Prospective Study to Compare the Impact on Motor, Neuropsychological, Psychiatric Outcomes and Quality of Life of STN-DBS Between Early Treated and Late-treated PD Patients.
Brief Title: Prospective Study to Compare Results of STN-DBS Between Early Treated and Late-treated PD Patient
Acronym: DeBraStE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: A.O. Ospedale Papa Giovanni XXIII (Other)
Collaborators: Associazione Italiana Parkinsoniani (AIP)- Sezione Bergamo (Unknown)
Responsible Party: Bruno Ferraro, Azienda Ospedaliera Ospedali Riuniti di Bergamo
Other Study IDs: BG200911
Record Dates: First submitted 2011-01-11; First posted 2011-01-12 (Estimated); Last update posted 2011-01-14 (Estimated); Status verified 2008-10

CONDITIONS: Parkinson's Disease; DBS; Deep Brain Stimulation; STN
Keywords: Parkinson; DBS of STN; PD; Deep Brain stimulation of STN; Early treatment
MeSH Terms: conditions — Parkinson Disease | interventions — Deep Brain Stimulation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Late-treated PD patients: Patients affected by Parkinson Disease, implanted with STN DBS and with an history of disease > 10 years
  Interventions: Device: Deep Brain Stimulation
- Early-treated PD patients: Patients affected by Parkinson Disease, implanted with STN DBS and with an history of disease <7 years
  Interventions: Device: Deep Brain Stimulation

INTERVENTIONS:
Device: Deep Brain Stimulation — Deep Brain Stimulation of STN in Parkinsonian patients
  Other Names: DBS

SUMMARY:
The aim of this study is to investigate the impact of DBS not only no motor outcomes, but also on neuropsychological and psychiatric aspects and on quality of life in young patients with a short history of disease.

DETAILED DESCRIPTION:
Bilateral STN DBS is a powerful treatment for advanced Parkinson disease with Levodopa induced motor complications. The beneficial effects of STN stimulation on motor disability and quality of life have been proved. However, the mean delay before neurosurgery is currently 14 years after diagnosis, when medical treatment no longer controls PD symptoms and quality of life is already severely impaired.

Aim of this study is to prospectively assess the effects of bilateral STN stimulation on motor signs, psychological and psychiatric aspects and quality of life in a group of 20 patients with PD who underwent surgery after 5 years from the onset of the disease. These results will be compared with those of a group of 20 patients with a PD history from more than 10 years.

The two groups of patients will be evaluated at baseline and after 3 and 12 months from DBS implant; at each visit neurological and motor examinations were assessed and dedicated neuropsychological and psychiatric tests will be performed.

Neurosurgery may be considered superior to medical treatment alone even in mild to moderate PD of 10 years duration, rather than a last resort in very advanced stages of the disease. Thanks to this study we could compare motor outcomes and cognitive aspects between DBS patients with a short and with long history of disease

ELIGIBILITY:
Inclusion Criteria:

* suffering from PD of > 10 years and with LTS (long term L-dopa syndrome), or with a duration of PD of 5 years
* age< 70 years
* normal brain MRI
* absence of dementia (Mini Mental State Examination ≥ 24)
* absence of severe psychiatric diseases
* Signed informed consent form
* Absence of allergy to metal
* Italian native speaker
* Absence of communicative or perceptive deficits

Exclusion Criteria:

* Any form of familiar PD
* Presence of neoplasia
* Presence of HIV
* Presence of severe metabolic diseases
* Severe cardiac/respiratory/renal or hepatic diseases
* Ongoing treatment with immunodepressive/ immunomodulate drugs

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This prospective clinical study will enroll 40 patients affected by PD. Patients enrolled will be divided into two groups based on the duration of disease. The first group will be composed by patients with PD duration of 5, while the second group will be composed by patients with a duration of disease longer than 10 years.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2011-02; Primary Completion 2013-04 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
percentage of improvement in motor aspects | after 12 months of stimulation
  The primary objective of the study is calculates as:
  (UPDRS III 12 months - UPDRS III baseline)/UPDRS III baseline
  where UPDRS III 12 months means the score of this test in "medication off , stimulation on" condition at 12 months after implant, while UPDRS III baseline means the score of this test in "medication off " condition.

SECONDARY OUTCOMES:
Neuropsychological aspects | after 3 and12 months of stimulation
  Evaluation of changes in the
  * global cognitive efficiency
  * short tem memory
  * attention
  * logical/executive functions
  * abstract reasoning
  * verbal fluency tasks
  * visuospatial and visuoconstructional abilities
Psychiatrical aspects | after 3 and12 months of stimulation
  Evaluation of changes in depression assessed by the Beck Depression Inventory
Quality of Life | after 3 and12 months of stimulation
  Evaluation of changes in quality of life assessed by PDQ39
Medication intake | after 3 and12 months of stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Ferraro, MD, Principal Investigator — Azienda Ospedaliera Ospedali Riuniti di Bergamo
Locations (1):
- Azienda Ospedaliera Ospedali Riuniti di Bergamo, Bergamo, Lombardy, Italy

REFERENCES:
- [Background] Lang AE, Lozano AM. Parkinson's disease. First of two parts. N Engl J Med. 1998 Oct 8;339(15):1044-53. doi: 10.1056/NEJM199810083391506. No abstract available. PMID 9761807
- [Background] Schrag A, Quinn N. Dyskinesias and motor fluctuations in Parkinson's disease. A community-based study. Brain. 2000 Nov;123 ( Pt 11):2297-305. doi: 10.1093/brain/123.11.2297. PMID 11050029
- [Background] Kumar R, Lozano AM, Kim YJ, Hutchison WD, Sime E, Halket E, Lang AE. Double-blind evaluation of subthalamic nucleus deep brain stimulation in advanced Parkinson's disease. Neurology. 1998 Sep;51(3):850-5. doi: 10.1212/wnl.51.3.850. PMID 9748038
- [Background] Moro E, Scerrati M, Romito LM, Roselli R, Tonali P, Albanese A. Chronic subthalamic nucleus stimulation reduces medication requirements in Parkinson's disease. Neurology. 1999 Jul 13;53(1):85-90. doi: 10.1212/wnl.53.1.85. PMID 10408541
- [Background] Vingerhoets FJ, Villemure JG, Temperli P, Pollo C, Pralong E, Ghika J. Subthalamic DBS replaces levodopa in Parkinson's disease: two-year follow-up. Neurology. 2002 Feb 12;58(3):396-401. doi: 10.1212/wnl.58.3.396. PMID 11839838
- [Background] Deep-Brain Stimulation for Parkinson's Disease Study Group; Obeso JA, Olanow CW, Rodriguez-Oroz MC, Krack P, Kumar R, Lang AE. Deep-brain stimulation of the subthalamic nucleus or the pars interna of the globus pallidus in Parkinson's disease. N Engl J Med. 2001 Sep 27;345(13):956-63. doi: 10.1056/NEJMoa000827. PMID 11575287
- [Background] Houeto JL, Damier P, Bejjani PB, Staedler C, Bonnet AM, Arnulf I, Pidoux B, Dormont D, Cornu P, Agid Y. Subthalamic stimulation in Parkinson disease: a multidisciplinary approach. Arch Neurol. 2000 Apr;57(4):461-5. doi: 10.1001/archneur.57.4.461. PMID 10768618
- [Background] Mesnage V, Houeto JL, Welter ML, Agid Y, Pidoux B, Dormont D, Cornu P. Parkinson's disease: neurosurgery at an earlier stage? J Neurol Neurosurg Psychiatry. 2002 Dec;73(6):778-9. doi: 10.1136/jnnp.73.6.778. No abstract available. PMID 12438494
- [Background] Carlesimo GA, Caltagirone C, Gainotti G. The Mental Deterioration Battery: normative data, diagnostic reliability and qualitative analyses of cognitive impairment. The Group for the Standardization of the Mental Deterioration Battery. Eur Neurol. 1996;36(6):378-84. doi: 10.1159/000117297. PMID 8954307
- [Result] Volkmann J. Deep brain stimulation for the treatment of Parkinson's disease. J Clin Neurophysiol. 2004 Jan-Feb;21(1):6-17. doi: 10.1097/00004691-200401000-00003. PMID 15097290
- [Result] Diamond A, Jankovic J. The effect of deep brain stimulation on quality of life in movement disorders. J Neurol Neurosurg Psychiatry. 2005 Sep;76(9):1188-93. doi: 10.1136/jnnp.2005.065334. PMID 16107348
- [Result] Schupbach WM, Maltete D, Houeto JL, du Montcel ST, Mallet L, Welter ML, Gargiulo M, Behar C, Bonnet AM, Czernecki V, Pidoux B, Navarro S, Dormont D, Cornu P, Agid Y. Neurosurgery at an earlier stage of Parkinson disease: a randomized, controlled trial. Neurology. 2007 Jan 23;68(4):267-71. doi: 10.1212/01.wnl.0000250253.03919.fb. Epub 2006 Dec 6. PMID 17151341